CLINICAL TRIAL: NCT06735924
Title: Non Alcoholic Fatty Liver Disease and Endogenous Oxalate Synthesis
Brief Title: Influence of Metabolic Syndrome on Endogenous Oxalate Synthesis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kyle D. Wood, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB300002318-FLO; 1R03DK139235-01 (NIH); UAB (Other: UAB)
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: MASLD; Metabolic Dysfunction-Associated Steatotic Liver Disease
Keywords: oxalate synthesis; oxalate metabolism; MASLD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Estimation of endogenous oxalate production (Experimental): Fasted hourly urine collections after equilibration on a low-oxalate diet
  Interventions: Dietary Supplement: Low-oxalate fixed diet

INTERVENTIONS:
Dietary Supplement: Low-oxalate fixed diet — Ingestion of a low-oxalate (< 60 mg/day) , normal calcium (800-1200 mg/d) eucaloric diet for 5 days

SUMMARY:
This study aims to determine the daily rate of endogenous synthesis of oxalate using fasted urine collection and a low-oxalate controlled diet in patients with Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD).

DETAILED DESCRIPTION:
Urinary oxalate excretion is derived from both dietary sources and endogenous synthesis. This study will use a low-oxalate controlled diet, repeat fasted urine collections and 24-hr urine collections on a low-oxalate diet, to determine the daily rate of endogenous oxalate synthesis in individuals with Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD).

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* History of MASLD, with liver fat content > 5%
* Normal kidney function
* Stable medication for at least 1 month for diabetes mellitus if any
* Willingess to ingest fixed diets and stop dietary supplements for the study and come to UAB for visits

Exclusion Criteria:

* Age < 18 years
* Inaccurate 24-hour urine collections
* Liver fat content <5%
* Liver cirrhosis
* Evidence of other chronic liver disease, viral hepatitis
* history of alcoholism within 2 years of enrollment
* Contra-indication to Magnetic Resonance Imaging
* Chronic kidney disease with estimated Glomerular Filtration rate < 60 ml/min/1.73m2
* Type 1 Diabetes Mellitus or treatment with insulin
* Uncontrolled diabetes
* Pregnancy, lactation or intention to be
* Uncontrolled hypertension
* Use of weight loss medication, SGLT2 inhibitors, GLP-1 receptor agonists, osteoporosis medication, chronic NSAID
* History of gastric or intestinal surgery or resection that could potentially alter oxalate absorption
* Chronic fat malabsorption
* Use of immunosuppressive medications
* Known immuno-compromised status
* Active malignancy or treatment for malignanacy within the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
estimated endogenous oxalate synthesis rate | 1 day
  Average fasted hourly urinary oxalate excretion rate normalized to urinary creatinine excretion (mg oxalate / g urinary creatinine)

SECONDARY OUTCOMES:
Urinary Oxalate excretion | 2 days
  average urinary oxalate excretion rate normalized to urinary creatinine after equilibration on a low-oxalate fixed diet (mg urinary oxalate / g urinary creatinine)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle D Wood, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No